CLINICAL TRIAL: NCT05343052
Title: Hamstring Injury (HAMIR) Index: A Framework for Injury Mitigations Strategies Through Innovative Imaging, Biomechanics, and Data Analytics
Brief Title: Hamstring Injury (HAMIR) Index
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Football League (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1420; A536130 (Other: UW Madison); Protocol Version 6/15/2023 (Other: UW Madison)
Record Dates: First submitted 2022-04-15; First posted 2022-04-25 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Hamstring Injury
Keywords: football; athlete
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Student Athlete: Student-athlete rostered on the varsity football team of participating institutions between 5/1/2022-6/30/2025 (study period)
  Interventions: Other: Patient Reported Outcomes Surveys; Other: Clinical Assessments; Other: Biomechanical and Neuromuscular Assessments; Device: Conventional MRI

INTERVENTIONS:
Other: Patient Reported Outcomes Surveys — * Oslo Sports Trauma Research Center Hamstring Injury Screening Questionnaire (HaOS) at baseline
  * Functional Assessment Scale for Acute Hamstring Injuries (FASH) within 7 days of injury and within 7 days of return to sport (RTS)
  Other Names: HaOS; FASH
Other: Clinical Assessments — * Injury History at baseline, within 7 days of injury, within 7 days of RTS
  * Pain and Function Assessments within 7 days of injury, within 7 days of RTS
Other: Biomechanical and Neuromuscular Assessments — * Eccentric Strength measure at baseline and within 7 days of RTS
  * Sprinting Biomechanics at baseline and within 7 days of RTS
Device: Conventional MRI — at baseline, within 7 days of injury, and within 7 days of RTS
  Other Names: Magnetic Resonance Imaging (MRI)

SUMMARY:
The investigators will combine state-of-the-art quantitative imaging, on-field biomechanics, and computational analytics into the largest-of-its-kind study to assess hamstring strain injury (HSI) risk and recovery in elite collegiate football players. The study will take place over 3 years and enroll up to 560 student athletes from Division I (D1) teams: University of Wisconsin-Madison, Brigham Young University and the University of North Carolina-Chapel Hill.

DETAILED DESCRIPTION:
The current approach to assess hamstring strain injury (HSI) risk and recovery is suboptimal. Many player-games are lost in American Football due to the lack of a clear understanding of the risk factors for HSI and the absence of effective methods to minimize re-injury.

The investigators propose that the key issues are: 1) every athlete is unique; therefore, a "one-size-fits-all" approach to HSI risk assessment will not work; 2) clinicians have limited relevant information on the potential injury risk for a specific athlete; 3) current methods to assess the extent of injury in a specific athlete are largely qualitative, limiting the ability to determine re-injury risk; and 4) current use of biologic injections is common, yet studies to quantify their effects are lacking. In this study, the investigators will address these four critical barriers by combining state-of-the-art quantitative imaging, on-field biomechanics, and computational analytics into the largest-of-its-kind study of elite collegiate football players.

The study will be conducted in 4 Division I collegiate men's football teams over a 3-year period. All student-athletes enrolled in this study will complete preseason hamstring strength testing, inertial measurement units (IMU)-based sprinting biomechanics, and undergo baseline magnetic resonance imaging (MRI). Student-athletes will be monitored by athletic trainers throughout the school year, who will record injuries and participation (e.g., time in practice, game).

Student-athletes who sustain an HSI will undergo a clinical assessment at the time of injury along with an MRI examination. Following completion of a rehabilitation program, hamstring strength will be re-evaluated and imaging will be repeated, along with performance measurements.

This study will provide the most detailed understanding of the physiological causes and effects of HSI, advancing our understanding of the processes affecting muscle function and improving our ability to evaluate, treat, and prevent HSI. This study represents what will be the largest, most quantitative prospective cohort study ever into HSI. Data gathered as part of this study will be used to develop a quantitative Hamstring Injury (HAMIR) index such that the medical and scientific communities can identify an individual athlete's propensity for HSI, and, more importantly, identify targets for injury mitigation, thereby reducing the global burden of HSI.

Aim 1. Develop a risk prediction model for HSI based on morphological, architectural, biomechanical and clinical factors in National Collegiate Athletic Association (NCAA) D1 college football players. The goal is to test the predictive capacity of innovative measures of risk for initial HSI in the largest prospective cohort study ever conducted in HSI. The outcome will be the establishment of a quantitative HAMIR index that is based on multiple athlete-specific measures. This aim will also identify potential future targets for injury risk mitigation and prophylactic strategies.

Aim 2. Develop a risk prediction model for recurrent HSI based on morphological, architectural, biomechanical and clinical factors (identified in Aim 1) in NCAA D1 college football players by completing the largest ever analysis of re-injury data. The investigators will track players who sustain an HSI, both immediately after injury and longitudinally. Quantification of injury metrics (e.g., volume of initial edema and volume, shape and location of long-term scar) will be incorporated into the analytics framework to develop a new "re-injury" HAMIR index. Similar to Aim 1, this aim will identify potential future targets for re-injury risk mitigation and prophylactic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Student-athlete rostered on the varsity football team of participating institutions between 5/1/2022-6/30/2025 (study period)

Exclusion Criteria:

* History of malignant disease
* Contraindication to MRI

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Student-athlete rostered on the varsity football team of participating institutions between 5/1/2022-6/30/2025 (study period)
Sampling Method: Non-Probability Sample
Enrollment: 699 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Aim 1: Initial Hamstring Strain Injury (HSI) | up to 3 years
  The outcome will be occurrence of an index HSI, measured at the athlete level. Athlete characteristics will be used to develop the quantitative HAMIR index to predict those at greatest risk of HSI. This aim will also identify potential future targets for injury risk mitigation and prophylactic strategies.
  HSI defined as an acute injury to the posterior thigh that limits full, unrestricted sports participation and includes two or more of the following symptoms: palpable pain along the hamstring muscles, posterior thigh pain without radicular symptoms, weakness and/or pain with resisted knee flexion, and pain with running.
Aim 2: Recurrent Hamstring Strain Injury (HSI) | up to 3 years
  The outcome will be the occurrence of a recurrent, or secondary, HSI measured at the athlete level. The investigators will use quantification of injury metrics (e.g., volume of initial edema and volume, shape and location of long-term scar) and incorporate these into the analytics framework to develop a new "re-injury" HAMIR index. Similar to Aim 1, this aim will identify potential future targets for re-injury risk mitigation and prophylactic approaches.
  Re-injury will be defined as an acute HSI that occurs to either limb within 6 months of an index HSI.

OTHER OUTCOMES:
Change in inertial measurement units (IMU)-based sprinting biomechanics | baseline and within 7 days of RTS (variable time points during training and within season)
  Sprinting biomechanics will be assessed using seven IMUs (sacrum, both thighs, both shanks, both feet). Lower extremity joint motions referenced to upright stance will be calculated throughout an on-field sprint and other football drills. After the completion of the running trial, onboard data from the IMUs will be downloaded and sent directly to Australian Catholic University from each site for further analysis.
Change in eccentric strength | baseline and within 7 days of RTS (variable time points during training and within season)
  Eccentric hamstring strength of each limb will be assessed during the Nordic hamstring exercise.
Change in Hamstring Outcome Score (HaOS) | baseline
  The HaOS is a functional patient reported outcome survey specific to their hamstring history (e.g. prior HSI) and hamstring function in training, competition and daily life. Scored on a 5 point likert scale from 0 (best score) to 4 (worst score). Sub-scores are calculated for each of the five main categories "Symptoms", "Soreness", "Pain", "Function, daily living and sports" and "Quality of life". The score is calculated in percent of the maximum score in each category, i.e. players without any complaints/symptoms would score 100 on each category. The total score is calculated as the mean of the five subscore percentages.
Change in Conventional MRI | baseline, within 7 days of injury, within 7 days of RTS (variable time points during training and within season)
  An MRI examination of the bilateral thighs will be performed on all student-athletes prior to the start of preseason (baseline) and repeated on those student-athletes that sustain an HSI at the time of injury and at time of return to sport. Coded MRIs will be sent directly to Springbok Analytics from each site, who will then be responsible for segmentation and analysis.
Change in Functional Assessment Scale for Acute Hamstring Injuries (FASH) Score | within 7 days of injury, within 7 days of RTS (variable time points during training and within season)
  The FASH is a 10-item assessment with a total possible range of scores from 0-100 where higher scores indicate better function.
Number of practice and competition exposures for each athlete | up to 3 years
  Athletic trainers will record weekly team reports that include the number of practice and competition exposures for each athlete. An injury risk exposure will be defined as one athlete participating in one practice or competition
Clinical Assessment of Pain | time of injury, within 7 days of RTS
  Location and length of pain via palpation. The location of maximum pain, as identified by the athlete, will be measured in centimeters from the ischial tuberosity. From the point of maximum pain, the hamstring will be palpated proximally and distally to determine the total length of pain, also measured in centimeters.
Functional Assessment: Range of Motion | time of injury, within 7 days of RTS
  Measured with goniometer to record full range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Heiderscheit, PT, PhD, FAPTA, Principal Investigator — UW School of Medicine and Public Health; David Opar, PhD, Principal Investigator — Australian Catholic University; Silvia Blemker, PhD, Principal Investigator — Springbok Analytics
Locations (5):
- United States (5):
  - Indiana University, Bloomington, Indiana
  - Notre Dame University, Notre Dame, Indiana
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Brigham Young University, Provo, Utah
  - University of Wisconsin - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heiderscheit BC, Blemker SS, Opar D, Stiffler-Joachim MR, Bedi A, Hart J, Mortensen B, Kliethermes SA; HAMIR Study Group. The development of a HAMstring InjuRy (HAMIR) index to mitigate injury risk through innovative imaging, biomechanics, and data analytics: protocol for an observational cohort study. BMC Sports Sci Med Rehabil. 2022 Jul 15;14(1):128. doi: 10.1186/s13102-022-00520-3. PMID 35841053